CLINICAL TRIAL: NCT06827145
Title: An Open-label, Single-center, Single-arm Phase IIa Study to Evaluate the Safety and Efficacy of Vebreltinib in Combination with Osimertinib in Patients with Locally Advanced or Metastatic Non-small Cell Lung Cancer with EGFR 21 L858R Mutation
Brief Title: Combination of Vebreltinib and Osimertinib in Patients with EGFR 21 L858R Mutation Advanced NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, China (Other)
Collaborators: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Puyuan Xing, Doctorate, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4728
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NSCLC; EGFR; Vebreltinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): All patients received oral Vebreltinib 100mg BID plus Osimertinib 80mg once daily.
  Interventions: Drug: Vebreltinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Vebreltinib — Vebreltinib 100mg oral BID
  Other Names: PLB1001; Bozitinib
Drug: Osimertinib — Osimertinib 80mg oral once daily.

SUMMARY:
This is a Prospective, open label, single arm study to evaluate the efficacy and safety of Vebreltinib combined with Osimertinib in the treatment of locally advanced or metastatic non-small cell lung cancer with EGFR 21 L858R mutation

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed an informed consent form.

  2. Patients aged ≥18.

  3. Histologically or cytologically confirmed locally or metastatic NSCLC.

  4.EGFR 21 L858R mutation.

  5.at least one measurable lesion according to RECIST 1.1 criteria.

  6.ECOG PS 0-1.

  7.appropriate organ function.

  8.For female subjects of reproductive age, a urine or serum pregnancy test should be performed negative within 7 days prior to receiving the first study drug administration .If there is a risk of conception, all subjects (male or female) must agree to use effective contraception from the time they sign an informed consent until 3 months after the final administration of the study drug.

  9.The expected survival is more than 3 months.

Exclusion Criteria:

* 1.Patients with EGFR 19del mutation , ALK or ROS1 gene fusions.

  2. Patients with symptomatic, neurologically unstable central nervous system (CNS) metastases, or CNS diseases that require increased steroid doses to control.

  3. Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.

  4.Previous treatment history meets one of the following criteria: 1)prior treated with systemic treatment. 2)The last administration of other anti-tumor drugs was less than 14 days or 5 half-life period before the initiation of study agents. 3)Received traditional Chinese medicine with anti-tumor indications within 1 week prior to initiation of treatment, 4)Thoracic radiotherapy to lung fields (including whole brain radiotherapy) ≤4 weeks prior to initiation of study treatment , for all other sites (except lung and whole brain) ≤2 weeks prior to initiation of study treatment. 5)Received major surgery within the past 4 weeks, or received resection of brain metastatic lesion within 2 weeks, or the side effects of such surgery have not yet been recovered.

  5.Previous anti-tumor therapy toxicity have not been recovered to ≤ Grade 1 (NCI-CTCAE 5.0) or baseline, except for alopecia, skin pigmentation and grade 2 peripheral neurotoxicity.

  6.Receive a potent inducer and/or potent inhibitor of CYP3A4 within 1 week prior to initiation of study drug or need receive a potent inducer and/or potent inhibitor of CYP3A4 during the study period.

  7.Any serious or uncontrolled systemic disease, including, but not limited to, other serious or psychiatric disorders or laboratory abnormalities, in which the investigator determines that the study drug is not suitable for the patient or affects protocol adherence.

  8.Cardiac function and disease meet one of the following criterias: QTc > 470 ms, Severe cardiac arrhythmia; Any risk factors that increase the length of the QTc; New York College of Cardiology (NYHA) Heart function grade ≥3. Poorly controlled hypertension.

  9.Have a history of interstitial lung disease, drug-induced interstitial lung disease, or radiation pneumonia requiring steroid therapy, or are currently receiving drug therapy or other clinical interventions, or have existing active interstitial lung disease.

  10.A history of thromboembolic or venous thromboembolic events (including myocardial infarction, cerebrovascular event or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other severe thromboembolic event) in the 6 months prior to the initial study drug administration, Any life-threatening bleeding event (including treatment requiring blood transfusion, surgery or local treatment, and ongoing medication) was judged to have a bleeding tendency.

  11.Active gastrointestinal disorders (such as ulcerative lesions, uncontrolled nausea, vomiting, diarrhea, and malabsorption syndrome) or other conditions (such as inability to swallow the investigational agent, or prior major gastrointestinal surgery) may significantly affect the absorption, distribution, metabolism, or excretion of the oral investigational agent.

  12.Patients with poorly controlled pleural effusion, peritoneal effusion, or pericardial effusion were judged by the investigators to be unsuitable for inclusion.

  13.Any systemic disease that the investigator determines to require treatment .

  14.A history of acute or chronic pancreatitis, pancreatic surgery, or risk factors that may increase the risk of developing pancreatitis.

  15.Active infection, including but not limited to:infected with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) (HIV antibody positive), infected with syphilis, active tuberculosis, the presence of active infections (such as pneumonia) requiring systematic anti-infective therapy within 2 weeks before drug administration in the first study.

  16.Patients being treated with warfarin or any other anticoagulant, except low-dose warfarin (< 2 mg) for the prevention of central catheter-associated thrombosis;

  17.Participants with known hypersensitivity or contraindications to study drug of same class or any excipient of these agents.

  18.Pregnant or lactating women.

  19.Patients were currently enrolled in another clinical study or received another clinical study drug within 2 weeks prior to initiation of study treatment.

  20. Other circumstances that, in the judgment of the investigator, may affect the conduct of the clinical study and the determination of the results of the study or increase the risks associated with drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  From the first treatment to the date of first documentation of disease progression, or death due to any cause

SECONDARY OUTCOMES:
Overall Response Rate | 3 years
  ORR is defined as the proportion of subjects with confirmed best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.
Overall survival | 5 years
  From the first administration to death from any cause
Duration of Response | 3 years
  DoR is defined as the time from the date of first documented response until date of documented progression per RECIST 1.1 as assessed by the investigator or death in the absence of disease progression.
Incidence of Treatment-Emergent Adverse Events | 3 years
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer insititue and Hospital of CHINESE ACADEMY OF MEDICAL SCIENCE, Beijing, China

IPD SHARING:
Plan to Share IPD: No